CLINICAL TRIAL: NCT05071768
Title: Focused ACT in Primary Care: A Pilot Study of a Virtual Group-based Intervention
Brief Title: Virtual Focused ACT Groups in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Erin Johns, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2021:298
Record Dates: First submitted 2021-09-15; First posted 2021-10-08 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Depression; Anxiety; Quality of Life; Acceptance Processes
MeSH Terms: conditions — Depression; Anxiety Disorders; Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT (Experimental): Focused ACT Group Treatment
  Interventions: Behavioral: Focused ACT

INTERVENTIONS:
Behavioral: Focused ACT — Brief acceptance and commitment therapy

SUMMARY:
Acceptance and commitment therapy (ACT) is a transdiagnostic intervention whose aim is to reduce experiential avoidance and promote psychological flexibility, which involves engaging in values-based behaviour while accepting painful internal experiences with openness and awareness. A growing body of research supports the efficacy of brief ACT for a variety of issues, including depression, anxiety, chronic pain, and stress. Given that ACT is a transdiagnostic intervention that targets the core processes related to human suffering, this treatment may be particularly useful for implementation in primary care with diverse groups of individuals and presentations. The objective of this study is to develop and pilot test a brief, virtual, group-based ACT intervention for depression and anxiety delivered in primary care settings to determine if a future randomized controlled trial of this group treatment is both warranted and feasible. The investigators will examine (1) the feasibility and acceptability of the study procedures, (2) clinician adherence to the treatment protocol, and (3) a preliminary analysis of the treatment effectiveness. A total of 3 groups (N = 30-45) will be conducted via three primary care clinics in Winnipeg, Manitoba, Canada. The group treatment will be delivered over four 90-minute sessions. Participants will complete assessment measures at pretreatment, post-treatment, and at two follow-up time points (1-month post-treatment and 3-6-months post-treatment). All assessments and treatment sessions will be conducted virtually via videoconferencing platform.

ELIGIBILITY:
Inclusion Criteria:

* self-reported symptoms of depression and/or anxiety
* fluent in English
* access to reliable internet and a device with a webcam as well as a private/quite space from which to attend sessions
* no change in psychotropic medication for at least 6 weeks prior to the intervention
* willingness to maintain a stable medication type and dose for psychotropic medications during the intervention phase and for one month post-intervention

Exclusion Criteria:

* engagement in another psychological treatment during the intervention phase or one month post-intervention
* current psychosis
* bipolar disorder
* current substance use disorder
* cognitive/intellectual impairment
* current active suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale 21-Items | Pretreatment
  21 items measuring depression, anxiety, and stress in the past week. Scores range from 0-42 for each of 3 scales (Depression, Anxiety, and Stress). Higher scores indicate worse outcomes (greater severity of depression, anxiety, and stress symptoms).
Depression Anxiety and Stress Scale 21-Items | 1 week following last treatment session
  21 items measuring depression, anxiety, and stress in the past week. Scores range from 0-42 for each of 3 scales (Depression, Anxiety, and Stress). Higher scores indicate worse outcomes (greater severity of depression, anxiety, and stress symptoms).
Depression Anxiety and Stress Scale 21-Items | 1-month follow-up
  21 items measuring depression, anxiety, and stress in the past week. Scores range from 0-42 for each of 3 scales (Depression, Anxiety, and Stress). Higher scores indicate worse outcomes (greater severity of depression, anxiety, and stress symptoms).
Depression Anxiety and Stress Scale 21-Items | 3-6-month follow-up
  21 items measuring depression, anxiety, and stress in the past week. Scores range from 0-42 for each of 3 scales (Depression, Anxiety, and Stress). Higher scores indicate worse outcomes (greater severity of depression, anxiety, and stress symptoms).
Acceptance and Action Questionnaire-II | Pretreament
  7 items measuring experiential avoidance. Scores range from 7-49. Higher scores indicate worse outcomes (less psychological flexibility).
Acceptance and Action Questionnaire-II | 1 week following last treatment session
  7 items measuring experiential avoidance. Scores range from 7-49. Higher scores indicate worse outcomes (less psychological flexibility).
Acceptance and Action Questionnaire-II | 1-month Follow-up
  7 items measuring experiential avoidance. Scores range from 7-49. Higher scores indicate worse outcomes (less psychological flexibility).
Acceptance and Action Questionnaire-II | 3-6-month Follow-up
  7 items measuring experiential avoidance. Scores range from 7-49. Higher scores indicate worse outcomes (less psychological flexibility).
Comprehensive assessment of Acceptance and Commitment Therapy processes | Pretreatment
  23 items measuring psychological flexibility (openness to experience, behavioural awareness, and valued action).
  Total score ranges from 0-138; higher scores indicate better outcomes (greater psychological flexibility).
  Openness to Experience subscale ranges from 0-60; higher scores indicate better outcomes (greater openness).
  Behavioural Awareness subscale ranges from 0-30; higher scores indicate better outcomes (greater behavioural awareness).
  Valued Action subscale ranges from 0-48; higher scores indicate better outcomes (greater valued action).
Comprehensive assessment of Acceptance and Commitment Therapy processes | 1 week following last treatment session
  23 items measuring psychological flexibility (openness to experience, behavioural awareness, and valued action).
  Total score ranges from 0-138; higher scores indicate better outcomes (greater psychological flexibility).
  Openness to Experience subscale ranges from 0-60; higher scores indicate better outcomes (greater openness).
  Behavioural Awareness subscale ranges from 0-30; higher scores indicate better outcomes (greater behavioural awareness).
  Valued Action subscale ranges from 0-48; higher scores indicate better outcomes (greater valued action).
Comprehensive assessment of Acceptance and Commitment Therapy processes | 1-month Follow-up
  23 items measuring psychological flexibility (openness to experience, behavioural awareness, and valued action).
  Total score ranges from 0-138; higher scores indicate better outcomes (greater psychological flexibility).
  Openness to Experience subscale ranges from 0-60; higher scores indicate better outcomes (greater openness).
  Behavioural Awareness subscale ranges from 0-30; higher scores indicate better outcomes (greater behavioural awareness).
  Valued Action subscale ranges from 0-48; higher scores indicate better outcomes (greater valued action).
Comprehensive assessment of Acceptance and Commitment Therapy processes | 3-6-month Follow-up
  23 items measuring psychological flexibility (openness to experience, behavioural awareness, and valued action).
  Total score ranges from 0-138; higher scores indicate better outcomes (greater psychological flexibility).
  Openness to Experience subscale ranges from 0-60; higher scores indicate better outcomes (greater openness).
  Behavioural Awareness subscale ranges from 0-30; higher scores indicate better outcomes (greater behavioural awareness).
  Valued Action subscale ranges from 0-48; higher scores indicate better outcomes (greater valued action).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Pretreatment
  16 items measuring level of satisfaction in different life domains (e.g., work, leisure activities, relationships).
  Scores range from 14-70. Higher scores indicate better outcomes (greater life satisfaction and enjoyment).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | 1 week following last treatment session
  16 items measuring level of satisfaction in different life domains (e.g., work, leisure activities, relationships).
  Scores range from 14-70. Higher scores indicate better outcomes (greater life satisfaction and enjoyment).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | 1-month Follow-up
  16 items measuring level of satisfaction in different life domains (e.g., work, leisure activities, relationships).
  Scores range from 14-70. Higher scores indicate better outcomes (greater life satisfaction and enjoyment).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | 3-6-month Follow-up
  16 items measuring level of satisfaction in different life domains (e.g., work, leisure activities, relationships).
  Scores range from 14-70. Higher scores indicate better outcomes (greater life satisfaction and enjoyment).

SECONDARY OUTCOMES:
Treatment Acceptability/Adherence Scale | Session 2 (2 weeks after start of treatment)
  10 items measuring treatment acceptability, adherence to treatment, and completion of treatment.
  Scores range from 10-70. Higher scores indicate better outcomes (greater treatment acceptability).
Percentage of planned treatment components delivered during treatment | Through treatment - 4 weeks
  Participant rating of whether planned treatment components were covered in each session Scores will be calculated as a percentage of agreement that planned topics were covered.
  Higher percentages indicate higher treatment integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Johns, PhD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - ACCESS Downtown, Winnipeg, Manitoba
  - ACCESS Winnipeg West, Winnipeg, Manitoba
  - ACCESS Fort Garry, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Coto-Lesmes R, Fernandez-Rodriguez C, Gonzalez-Fernandez S. Acceptance and Commitment Therapy in group format for anxiety and depression. A systematic review. J Affect Disord. 2020 Feb 15;263:107-120. doi: 10.1016/j.jad.2019.11.154. Epub 2019 Dec 2. PMID 31818766
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Schechter D, Endicott J, Nee J. Quality of life of 'normal' controls: association with lifetime history of mental illness. Psychiatry Res. 2007 Jul 30;152(1):45-54. doi: 10.1016/j.psychres.2006.09.008. Epub 2007 Mar 23. PMID 17363070